CLINICAL TRIAL: NCT02684903
Title: Coaching Alternative Parenting Strategies (CAPS) Study: Targeting Neurobiological and Behavioral Mechanisms of Self-regulation in High-risk Families
Brief Title: Coaching Alternative Parenting Strategies (CAPS) Study
Acronym: CAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Principal Investigator, Elizabeth Skowron, Professor, Department of Psychology, University of Oregon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01DA036533-01A1 (NIH)
Record Dates: First submitted 2016-02-02; First posted 2016-02-18 (Estimated); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Child Abuse; Self-control; Parenting
Keywords: Child Abuse; Parent Child Interaction Therapy (PCIT); Evidenced Based Intervention; Self-control
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Services As Usual (SAU) (No Intervention): Participants receive all the usual services provided by Department of Human Services (DHS) Children's Services.
- Parent Child Interaction Therapy (PCIT) (Experimental): Participants receive Parent Child Interaction Therapy (PCIT). PCIT is designed to improve child functioning by interrupting patterns of harsh, coercive interaction and enhancing parents' warm, positive parenting, autonomy support, and competent child management skills.
  .
  Interventions: Behavioral: Parent Child Interaction Therapy

INTERVENTIONS:
Behavioral: Parent Child Interaction Therapy — PCIT is a 16-20 session live-coaching parenting intervention. PCIT for Child Welfare families is delivered in two sequential treatment phases following a motivational enhancement training: Phase 1, Child-Directed Interaction (CDI) to enhance positive parenting and interrupt harsh aversive parenting, and Phase 2, Parent-Directed Interaction (PDI) to coach effective parent commands and a consistent time-out protocol when child disobeys.
  Other Names: PCIT
  Arms: Parent Child Interaction Therapy (PCIT)

SUMMARY:
This is a randomized, controlled trial (RCT) of Parent-Child Interaction Therapy (PCIT) designed to test the effects of PCIT on self-regulation and behavior in child maltreating (CM) parents and their elementary-school children. Two hundred-fifty (250) maltreating mothers and their children (age 5-8 years) will be drawn from Child Protective Services and randomized to the PCIT intervention or a control condition (services as usual). Key contextual risk factors will be assessed, including cumulative risk, parent mental health, and parent substance use. A multirater, multimethod approach to assessment will include measures of self-regulation, parenting skills and children's behavior outcomes. Families will be followed to 1 year for CM recidivism. Findings from this proposed study are expected to have significant implications for optimizing CM parenting interventions by (a) determining the sensitivity of CM parent and child neurobehavioral self-regulation systems to intervention, and (b) identifying individual differences in self-regulation that mediate and moderate response to intervention and long-term maintenance of gains.

DETAILED DESCRIPTION:
Child maltreatment (CM) constitutes a serious public health problem in the United States and is known to compromise children's developing self-regulation skills and amplify risk for substance use and other regulatory disorders. Parent-Child Interaction Therapy (PCIT), an intensive, 20-session parenting intervention, has been shown to improve the quality of CM parenting, improve positive parenting and child behavior, and produce declines in CM recidivism (Chaffin et al., 2004) though the mechanisms underlying its effects are little understood. This project addresses gaps in the CM intervention literature in that it (a) uses an experimental intervention design to test a theoretical model of change underlying PCIT's effects, (b) includes a battery of neurobehavioral measures of self-regulation, and (c) uses observational measures of parenting in an RCT of an evidence-based intervention for strengthening parent self-regulation, reducing CM, and supporting improvements in child regulation and behavior. Study aims are to:

Aim 1: Test the main effects of PCIT on CM-specific outcomes, including reductions in harsh, aversive parenting and CM recidivism and promotion of children's behavioral adjustment. It is hypothesized that intervention families will show significantly greater behavior improvements (i.e., decreased negative parenting, increased positive parenting, and decreased child internalizing/externalizing problems) at posttest and lower CM recidivism at 6-month follow-up, compared to families receiving services as usual (SAU).

Specific Aim 2: Determine the impact of PCIT on indices of CM parents' self-regulation. First, the investigators will test the hypothesis that PCIT exerts direct effects on improving CM parents' capacities for self-regulation in the context of parenting. Second, the investigators will investigate how measures of self-regulation in parents mediate PCIT intervention effects on reductions in CM and improvements in parenting. Third, the investigators will explore whether parents' preintervention self-regulation levels moderate intervention effects on outcomes. The moderating roles of CM subtype (i.e., physical abuse vs. neglect), severity, and other key sociocontextual factors on the outcomes of interest also will be considered.

Specific Aim 3: Investigate the impact of PCIT on neurobehavioral indices of CM children's self-regulation. CM exerts detrimental effects on children's developing capacities to regulate attention, emotion, physiology, and behavior. Deficits in these domains confer heightened risk for psychopathology, early-onset conduct problems, and later substance abuse. The investigators hypothesize that PCIT, though directed primarily toward parenting, will effect improvements in neurobiological indicators of CM children's self-regulation at post-treatment, relative to the control group. Next, the investigators will test the extent to which child outcomes are mediated through intervention effects on parenting. It is hypothesized that child regulatory deficits and behavior problems will be attenuated by PCIT-based reductions in aversive parenting that result from the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Lane County
* Parent is 18 or older
* Biological or custodial mother of a child between age 3 and 7 years at baseline
* Resides in the same home setting with the child
* Must be fluent in English
* Mom and child must be physically able to complete the assessment
* Family has an open case with Lane County Dept. Health Services.

Exclusion Criteria:

* Child sexual abuse in the family

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2022-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Skowron, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

REFERENCES:
- [Background] Aber JL, Cicchetti D. The social-emotional development of maltreated children: An empirical and theoretical analysis. In H. Fitzgerald, B. Lester, & M. Yogman (Eds.), Theory and research in behavioral pediatrics (Vol. 2, pp. 147-205). New York, NY: Plenum, 1984.
- [Background] Abidin RR. Parenting Stress Index (3rd ed.). Odessa, FL: Psychological Assessment Resources, 1995.
- [Background] Achenbach TM, Rescorla LA. Manual for the ASEBA School-Age Forms and Profiles. Burlington, VT: University of Vermont, Research Center for Children, Youth, and Families, 2001.
- [Background] Adler NE, Epel ES, Castellazzo G, Ickovics JR. Relationship of subjective and objective social status with psychological and physiological functioning: preliminary data in healthy white women. Health Psychol. 2000 Nov;19(6):586-92. doi: 10.1037//0278-6133.19.6.586. PMID 11129362
- [Background] Alkon A, Goldstein LH, Smider N, Essex MJ, Kupfer DJ, Boyce WT. Developmental and contextual influences on autonomic reactivity in young children. Dev Psychobiol. 2003 Jan;42(1):64-78. doi: 10.1002/dev.10082. PMID 12471637
- [Background] Anderson TW, Amemiya Y. The asymptotic normal distribution of estimators in factor analysis under general conditions. The Annals of Statistics 16(2): 759-771, 1988.
- [Background] Aos S, Lee S, Drake E, Pennucci A, Klima T, Miller M, Anderson L, Mayfield J, Burley M. Return on investment: Evidence-based options to improve statewide outcomes (Document No. 11-07-1201). Olympia: Washington State Institute for Public Policy, 2011.
- [Background] Barnett D, Manly JT, Cicchetti D. Defining child maltreatment: The interface between policy and research. In D. Cicchetti & S. L. Toth (Eds.), Child abuse, child development, and social policy (pp. 7-73). Norwood, NJ: Ablex, 1993.
- [Background] Bäumler G.Farb-Wort-Interferenztest (FWIT) nach J.R. Stroop. Göttingen: Hogrefe, 1985.
- [Background] Beauchaine T. Vagal tone, development, and Gray's motivational theory: toward an integrated model of autonomic nervous system functioning in psychopathology. Dev Psychopathol. 2001 Spring;13(2):183-214. doi: 10.1017/s0954579401002012. PMID 11393643
- [Background] Beauchaine TP, Gatzke-Kopp L, Mead HK. Polyvagal Theory and developmental psychopathology: emotion dysregulation and conduct problems from preschool to adolescence. Biol Psychol. 2007 Feb;74(2):174-84. doi: 10.1016/j.biopsycho.2005.08.008. Epub 2006 Oct 12. PMID 17045726
- [Background] Beauchaine TP, Neuhaus E, Brenner SL, Gatzke-Kopp L. Ten good reasons to consider biological processes in prevention and intervention research. Dev Psychopathol. 2008 Summer;20(3):745-74. doi: 10.1017/S0954579408000369. PMID 18606030
- [Background] Beckett LA, Tancredi DJ, Wilson RS. Multivariate longitudinal models for complex change processes. Stat Med. 2004 Jan 30;23(2):231-9. doi: 10.1002/sim.1712. PMID 14716725
- [Background] Belsky J. Etiology of child maltreatment: a developmental-ecological analysis. Psychol Bull. 1993 Nov;114(3):413-34. doi: 10.1037/0033-2909.114.3.413. PMID 8272464
- [Background] Berger A. Neurocognitive and neuromotivational mechanisms of self-regulation. In A. Berger (Ed.), Self-regulation: Brain, cognition, and development. Human brain development series, (pp. 19-44). Washington, DC: American Psychological Association, 2011.
- [Background] Berkman ET, Kahn LE, Merchant JS. Training-induced changes in inhibitory control network activity. J Neurosci. 2014 Jan 1;34(1):149-57. doi: 10.1523/JNEUROSCI.3564-13.2014. PMID 24381276
- [Background] Berliner L, Elliott DM. Sexual abuse of children. In J. E. B. Myers, L. Berliner, J. Briere, C. T. Hendrix, C. Jenny, & T. A. Reid (Eds.), The APSAC handbook on child maltreatment (2nd ed., pp. 55-78). Thousand Oaks, CA: Sage, 2002.
- [Background] Berntson GG, Bigger JT Jr, Eckberg DL, Grossman P, Kaufmann PG, Malik M, Nagaraja HN, Porges SW, Saul JP, Stone PH, van der Molen MW. Heart rate variability: origins, methods, and interpretive caveats. Psychophysiology. 1997 Nov;34(6):623-48. doi: 10.1111/j.1469-8986.1997.tb02140.x. PMID 9401419
- [Background] Berntson GG, Cacioppo JT, Quigley KS, Fabro VT. Autonomic space and psychophysiological response. Psychophysiology. 1994 Jan;31(1):44-61. doi: 10.1111/j.1469-8986.1994.tb01024.x. PMID 8146254
- [Background] Bierman KL, Nix RL, Greenberg MT, Blair C, Domitrovich CE. Executive functions and school readiness intervention: impact, moderation, and mediation in the Head Start REDI program. Dev Psychopathol. 2008 Summer;20(3):821-43. doi: 10.1017/S0954579408000394. PMID 18606033
- [Background] Bollen KA, Curran PJ. Latent curve models: A structural equation perspective. Hoboken, NJ: John Wiley & Sons, 2006.
- [Background] Borrego J, Timmer SG, Urquiza AJ, Follette WC. Physically abusive mothers' responses following episodes of child noncompliance and compliance. J Consult Clin Psychol. 2004 Oct;72(5):897-903. doi: 10.1037/0022-006X.72.5.897. PMID 15482048
- [Background] Briere J, Johnson K, Bissada A, Damon L, Crouch J, Gil E, Hanson R, Ernst V. The Trauma Symptom Checklist for Young Children (TSCYC): reliability and association with abuse exposure in a multi-site study. Child Abuse Negl. 2001 Aug;25(8):1001-14. doi: 10.1016/s0145-2134(01)00253-8. PMID 11601594
- [Background] Browne MW. Robustness of statistical inference in factor analysis and related models. Biometrika 74(2): 375-384, 1987.
- [Background] Bruce J, Fisher PA, Pears KC, Levine S. Morning cortisol Levels in preschool-aged foster children: differential effects of maltreatment type. Dev Psychobiol. 2009 Jan;51(1):14-23. doi: 10.1002/dev.20333. PMID 18720365
- [Background] Bruce J, McDermott JM, Fisher PA, Fox NA. Using behavioral and electrophysiological measures to assess the effects of a preventive intervention: a preliminary study with preschool-aged foster children. Prev Sci. 2009 Jun;10(2):129-40. doi: 10.1007/s11121-008-0115-8. PMID 19030992
- [Background] Bryck RL, Fisher PA. Training the brain: practical applications of neural plasticity from the intersection of cognitive neuroscience, developmental psychology, and prevention science. Am Psychol. 2012 Feb-Mar;67(2):87-100. doi: 10.1037/a0024657. Epub 2011 Jul 25. PMID 21787037
- [Background] Bryk AS, Raudenbush SW. Hierarchical linear models: Applications and data analysis methods. Newbury Park, CA: Sage, 1992.
- [Background] Bugental DB. Predicting & preventing child maltreatment: A biocognitive transactional approach. In A. Sameroff (Ed.), The transactional model of development: How children and contexts shape each other (pp. 97-115). Washington, DC: American Psychological Association, 2009.
- [Background] Bugental DB, Ellerson PC, Lin EK, Rainey B, Kokotovic A, O'Hara N. A cognitive approach to child abuse prevention. J Fam Psychol. 2002 Sep;16(3):243-58. doi: 10.1037//0893-3200.16.3.243. PMID 12238408
- [Background] Bush NR, Alkon A, Obradovic J, Stamperdahl J, Boyce WT. Differentiating challenge reactivity from psychomotor activity in studies of children's psychophysiology: considerations for theory and measurement. J Exp Child Psychol. 2011 Sep;110(1):62-79. doi: 10.1016/j.jecp.2011.03.004. Epub 2011 Apr 27. PMID 21524757
- [Background] Butler EA, Wilhelm FH, Gross JJ. Respiratory sinus arrhythmia, emotion, and emotion regulation during social interaction. Psychophysiology. 2006 Nov;43(6):612-22. doi: 10.1111/j.1469-8986.2006.00467.x. PMID 17076818
- [Background] Cacioppo JT, Uchino BN, Berntson GG. Individual differences in the autonomic origins of heart rate reactivity: the psychometrics of respiratory sinus arrhythmia and preejection period. Psychophysiology. 1994 Jul;31(4):412-9. doi: 10.1111/j.1469-8986.1994.tb02449.x. PMID 10690921
- [Background] Capage LC, Bennett GM, McNeil, CB. A comparison between African American and Caucasian children referred for treatment of disruptive behavior disorders. Child and Family Behavior Therapy. 23: 1-14, 2001.
- [Background] Carmichael-Olsen H, Greenberg MT, Slough N. Coding manual for the waiting task. Unpublished manual, University of Washington, Seattle, 1985.
- [Background] Chaffin M, Funderburk B, Bard D, Valle LA, Gurwitch R. A combined motivation and parent-child interaction therapy package reduces child welfare recidivism in a randomized dismantling field trial. J Consult Clin Psychol. 2011 Feb;79(1):84-95. doi: 10.1037/a0021227. PMID 21171738
- [Background] Chaffin M, Silovsky JF, Funderburk B, Valle LA, Brestan EV, Balachova T, Jackson S, Lensgraf J, Bonner BL. Parent-child interaction therapy with physically abusive parents: efficacy for reducing future abuse reports. J Consult Clin Psychol. 2004 Jun;72(3):500-510. doi: 10.1037/0022-006X.72.3.500. PMID 15279533
- [Background] Chaffin M, Valle LA, Funderburk B, Gurwitch R, Silovsky J, Bard D, McCoy C, Kees M. A motivational intervention can improve retention in PCIT for low-motivation child welfare clients. Child Maltreat. 2009 Nov;14(4):356-68. doi: 10.1177/1077559509332263. Epub 2009 Mar 2. PMID 19258303
- [Background] Chang L, Schwartz D, Dodge KA, McBride-Chang C. Harsh parenting in relation to child emotion regulation and aggression. J Fam Psychol. 2003 Dec;17(4):598-606. doi: 10.1037/0893-3200.17.4.598. PMID 14640808
- [Background] Chapman HA, Woltering S, Lamm C, Lewis MD. Hearts and minds: Coordination of neurocognitive and cardiovascular regulation in children and adolescents. Biol Psychol. 2010 May;84(2):296-303. doi: 10.1016/j.biopsycho.2010.03.001. Epub 2010 Mar 17. PMID 20223274
- [Background] Cicchetti D, Rizley R. Developmental perspectives on the etiology, intergenerational transmission, and sequelae of child maltreatment. New Directions for Child Development 11: 31-55, 1981.
- [Background] Cicchetti D, Toth SL. Child maltreatment. Annu Rev Clin Psychol. 2005;1:409-38. doi: 10.1146/annurev.clinpsy.1.102803.144029. PMID 17716094
- [Background] Cicchetti D, Rogosch FA, Gunnar MR, Toth SL. The differential impacts of early physical and sexual abuse and internalizing problems on daytime cortisol rhythm in school-aged children. Child Dev. 2010 Jan-Feb;81(1):252-69. doi: 10.1111/j.1467-8624.2009.01393.x. PMID 20331666
- [Background] Cicchetti D, Rogosch FA, Toth SL, Sturge-Apple ML. Normalizing the development of cortisol regulation in maltreated infants through preventive interventions. Dev Psychopathol. 2011 Aug;23(3):789-800. doi: 10.1017/S0954579411000307. PMID 21756432
- [Background] Cipriano EA, Skowron EA, Gatzke-Kopp LM. Preschool children's cardiac reactivity moderates relations between exposure to family violence and emotional adjustment. Child Maltreat. 2011 Aug;16(3):205-15. doi: 10.1177/1077559511408887. Epub 2011 May 17. PMID 21593016
- [Background] Cohen J. Statistical power analysis for the social sciences (2nd ed.). Hillsdale, NJ: Erlbaum, 1988.
- [Background] Conduct Problems Prevention Research Group (CPPRG). (1994). Financial Stress Questionnaire. Available from the Fast Track Project Web site, http://fasttrackproject.org
- [Background] Cowan PA, Cowan CP. Interventions as tests of family systems theories: marital and family relationships in children's development and psychopathology. Dev Psychopathol. 2002 Fall;14(4):731-59. doi: 10.1017/s0954579402004054. PMID 12549702
- [Background] Creaven AM, Skowron EA, Hughes BM, Howard S, Loken E. Dyadic concordance in mother and preschooler resting cardiovascular function varies by risk status. Dev Psychobiol. 2014 Jan;56(1):142-52. doi: 10.1002/dev.21098. Epub 2013 Sep 11. PMID 24022469
- [Background] Curtis WJ, Cicchetti D. Affective facial expression processing in young children who have experienced maltreatment during the first year of life: an event-related potential study. Dev Psychopathol. 2011 May;23(2):373-95. doi: 10.1017/S0954579411000125. PMID 23786684
- [Background] Dahl RE. Adolescent brain development: a period of vulnerabilities and opportunities. Keynote address. Ann N Y Acad Sci. 2004 Jun;1021:1-22. doi: 10.1196/annals.1308.001. PMID 15251869
- [Background] Davies PT, Cicchetti D. Toward an integration of family systems and developmental psychopathology approaches. Dev Psychopathol. 2004 Summer;16(3):477-81. doi: 10.1017/s0954579404004626. No abstract available. PMID 15605621
- [Background] De Bellis MD. The psychobiology of neglect. Child Maltreat. 2005 May;10(2):150-72. doi: 10.1177/1077559505275116. PMID 15798010
- [Background] Deater-Deckard K, Sewell MD, Petrill SA, Thompson LA. Maternal working memory and reactive negativity in parenting. Psychol Sci. 2010 Jan;21(1):75-9. doi: 10.1177/0956797609354073. Epub 2009 Nov 23. PMID 20424026
- [Background] Derogatis L. Brief Symptom Inventory (BSI): Administration, scoring, and procedures manual (3rd ed.). Minneapolis, MN: National Computer Systems, 1993.
- [Background] Dix T. The affective organization of parenting: adaptive and maladaptive processes. Psychol Bull. 1991 Jul;110(1):3-25. doi: 10.1037/0033-2909.110.1.3. PMID 1891517
- [Background] Dodge KA, Bates JE, Pettit GS. Mechanisms in the cycle of violence. Science. 1990 Dec 21;250(4988):1678-83. doi: 10.1126/science.2270481.
- [Background] Dozier M, Kobak RR. Psychophysiology in attachment interviews: converging evidence for deactivating strategies. Child Dev. 1992 Dec;63(6):1473-80. PMID 1446563
- [Background] Ellis BJ, Boyce WT, Belsky J, Bakermans-Kranenburg MJ, van Ijzendoorn MH. Differential susceptibility to the environment: an evolutionary--neurodevelopmental theory. Dev Psychopathol. 2011 Feb;23(1):7-28. doi: 10.1017/S0954579410000611. PMID 21262036
- [Background] Emery RE, Laumann-Billings L. An overview of the nature, causes, and consequences of abusive family relationships. Toward differentiating maltreatment and violence. Am Psychol. 1998 Feb;53(2):121-35. doi: 10.1037//0003-066x.53.2.121. PMID 9491743
- [Background] Enders CK. The impact of nonnormality on full information maximum-likelihood estimation for structural equation models with missing data. Psychol Methods. 2001 Dec;6(4):352-70. PMID 11778677
- [Background] Erickson MF, Egeland B, Pianta R. The effects of maltreatment on the development of young children. In D. Cicchetti & V. Carlson (Eds.), Child maltreatment: Theory and research on the causes and consequences of child abuse and neglect (pp. 647-684). New York, NY: Cambridge University Press, 1989.
- [Background] Evans GW, English K. The environment of poverty: multiple stressor exposure, psychophysiological stress, and socioemotional adjustment. Child Dev. 2002 Jul-Aug;73(4):1238-48. doi: 10.1111/1467-8624.00469. PMID 12146745
- [Background] Eyberg SM, Funderburk B. Parent-child interaction therapy protocol. Gainesville, FL: PCIT International, 2011.
- [Background] Eyberg SM, Pincus D. Eyberg Child Behavior Inventory & Sutter-Eyberg Student Behavior Inventory-Revised: Professional Manual. Odessa, FL: Psychological Assessment Resources, 1999.
- [Background] Eyberg SM, Funderburk BW, Hembree-Kigin TL, McNeil CB, Querido JG, Hood KK. Parent-Child Interaction Therapy with behavior problem children: One and two year maintenance of treatment effects in the family. Child & Family Behavior Therapy 23: 1-20, 2001.
- [Background] Robinson EA, Eyberg SM. The dyadic parent-child interaction coding system: standardization and validation. J Consult Clin Psychol. 1981 Apr;49(2):245-50. doi: 10.1037//0022-006x.49.2.245. No abstract available. PMID 7217491
- [Background] Falkenstein M, Hoormann J, Hohnsbein J. ERP components in Go/Nogo tasks and their relation to inhibition. Acta Psychol (Amst). 1999 Apr;101(2-3):267-91. doi: 10.1016/s0001-6918(99)00008-6. PMID 10344188
- [Background] Farver JA, Xu Y, Eppe S, Fernandez A, Schwartz D. Community violence, family conflict, and preschoolers' socioemotional functioning. Dev Psychol. 2005 Jan;41(1):160-70. doi: 10.1037/0012-1649.41.1.160. PMID 15656746
- [Background] Feil EG, Baggett KM, Davis B, Sheeber L, Landry S, Carta JJ, Buzhardt J. Expanding the reach of preventive interventions: development of an Internet-based training for parents of infants. Child Maltreat. 2008 Nov;13(4):334-46. doi: 10.1177/1077559508322446. PMID 18843143
- [Background] Fisher PA, Gunnar MR, Dozier M, Bruce J, Pears KC. Effects of therapeutic interventions for foster children on behavioral problems, caregiver attachment, and stress regulatory neural systems. Ann N Y Acad Sci. 2006 Dec;1094:215-25. doi: 10.1196/annals.1376.023. PMID 17347353
- [Background] Funderburk BW, Eyberg SM. History of parent-child interaction therapy. In J. Norcross (Ed.), History of Psychotherapy: Continuity and change (2nd ed., pp.415-420). Washington, DC: American Psychological Association, 2010.
- [Background] Gerstadt CL, Hong YJ, Diamond A. The relationship between cognition and action: performance of children 3 1/2-7 years old on a Stroop-like day-night test. Cognition. 1994 Nov;53(2):129-53. doi: 10.1016/0010-0277(94)90068-x. PMID 7805351
- [Background] Baron IS. Behavior rating inventory of executive function. Child Neuropsychol. 2000 Sep;6(3):235-8. doi: 10.1076/chin.6.3.235.3152. No abstract available. PMID 11419452
- [Background] Giuliano RJ, Skowron EA, Berkman ET. Growth models of dyadic synchrony and mother-child vagal tone in the context of parenting at-risk. Biol Psychol. 2015 Feb;105:29-36. doi: 10.1016/j.biopsycho.2014.12.009. Epub 2014 Dec 24. PMID 25542759
- [Background] Graziano P, Derefinko K. Cardiac vagal control and children's adaptive functioning: a meta-analysis. Biol Psychol. 2013 Sep;94(1):22-37. doi: 10.1016/j.biopsycho.2013.04.011. Epub 2013 May 4. PMID 23648264
- [Background] Graziano PA, Bagner DM, Sheinkopf SJ, Vohr BR, Lester BM. Evidence-based intervention for young children born premature: preliminary evidence for associated changes in physiological regulation. Infant Behav Dev. 2012 Jun;35(3):417-28. doi: 10.1016/j.infbeh.2012.04.001. Epub 2012 Jun 19. PMID 22721742
- [Background] Gresham FM, Elliott SN. Social Skills Improvement System Rating Scales manual. Minneapolis, MN: NCS Pearson, 2008.
- [Background] Gunnar MR, Fisher PA; Early Experience, Stress, and Prevention Network. Bringing basic research on early experience and stress neurobiology to bear on preventive interventions for neglected and maltreated children. Dev Psychopathol. 2006 Summer;18(3):651-77. PMID 17152395
- [Background] Gunnar M, Quevedo K. The neurobiology of stress and development. Annu Rev Psychol. 2007;58:145-73. doi: 10.1146/annurev.psych.58.110405.085605. PMID 16903808
- [Background] Hagger MS, Wood C, Stiff C, Chatzisarantis NL. Ego depletion and the strength model of self-control: a meta-analysis. Psychol Bull. 2010 Jul;136(4):495-525. doi: 10.1037/a0019486. PMID 20565167
- [Background] Hajcak G, Nieuwenhuis S. Reappraisal modulates the electrocortical response to unpleasant pictures. Cogn Affect Behav Neurosci. 2006 Dec;6(4):291-7. doi: 10.3758/cabn.6.4.291. PMID 17458444
- [Background] Hajcak G, MacNamara A, Olvet DM. Event-related potentials, emotion, and emotion regulation: an integrative review. Dev Neuropsychol. 2010;35(2):129-55. doi: 10.1080/87565640903526504. PMID 20390599
- [Background] Hakman M, Chaffin M, Funderburk B, Silovsky JF. Change trajectories for parent-child interaction sequences during parent-child interaction therapy for child physical abuse. Child Abuse Negl. 2009 Jul;33(7):461-70. doi: 10.1016/j.chiabu.2008.08.003. Epub 2009 Jul 5. PMID 19581001
- [Background] Heaton RK, & PAR Staff. Wisconsin Card Sorting Test: Computer version 4. Odessa, FL: Psychological Assessment Resources, 2003.
- [Background] Heller SS, Larrieu JA, D'Imperio R, Boris NW. Research on resilience to child maltreatment: empirical considerations. Child Abuse Negl. 1999 Apr;23(4):321-38. doi: 10.1016/s0145-2134(99)00007-1. PMID 10321770
- [Background] Hertsgaard L, Gunnar M, Erickson MF, Nachmias M. Adrenocortical responses to the strange situation in infants with disorganized/disoriented attachment relationships. Child Dev. 1995 Aug;66(4):1100-6. PMID 7671652
- [Background] Hoffman C, Crnic KA, Baker JK. Maternal depression and parenting: Implications for children's emergent emotion regulation and behavioral functioning. Parenting: Science and Practice 6: 271-295, 2006.
- [Background] Joosen KJ, Mesman J, Bakermans-Kranenburg MJ, van Ijzendoorn MH. Maternal overreactive sympathetic nervous system responses to repeated infant crying predicts risk for impulsive harsh discipline of infants. Child Maltreat. 2013 Nov;18(4):252-63. doi: 10.1177/1077559513494762. Epub 2013 Jul 8. PMID 23836807
- [Background] Judd CM, Kenny DA, McClelland GH. Estimating and testing mediation and moderation in within-subject designs. Psychol Methods. 2001 Jun;6(2):115-34. doi: 10.1037/1082-989x.6.2.115. PMID 11411437
- [Background] Kaufman J, Zigler, EF. The intergenerational transmission of child abuse. In D. Cicchetti & V. Carlson (Eds.), Child maltreatment: Theory and research on the causes and consequences of child abuse and neglect (pp. 129-150). New York, NY: Cambridge University Press, 1989.
- [Background] Kerr ME, Bowen M. Family evaluation. New York, NY: Norton, 1988.
- [Background] Knudsen DD. Child Protective Services: Discretion, decisions, dilemmas. Springfield, IL: Charles C. Thomas Publisher, 1988.
- [Background] Kopp CB. Regulation of distress and negative emotions: A developmental review. Developmental Psychology 25: 343-354, 1989.
- [Background] Loeber R, Hay D. Key issues in the development of aggression and violence from childhood to early adulthood. Annu Rev Psychol. 1997;48:371-410. doi: 10.1146/annurev.psych.48.1.371. PMID 9046564
- [Background] Loman MM, Johnson AE, Westerlund A, Pollak SD, Nelson CA, Gunnar MR. The effect of early deprivation on executive attention in middle childhood. J Child Psychol Psychiatry. 2013 Jan;54(1):37-45. doi: 10.1111/j.1469-7610.2012.02602.x. Epub 2012 Aug 24. PMID 22924462
- [Background] MacKinnon DP, Luecken LJ. How and for whom? Mediation and moderation in health psychology. Health Psychol. 2008 Mar;27(2S):S99-S100. doi: 10.1037/0278-6133.27.2(Suppl.).S99. PMID 18377161
- [Background] MacKinnon DP, Fritz MS, Williams J, Lockwood CM. Distribution of the product confidence limits for the indirect effect: program PRODCLIN. Behav Res Methods. 2007 Aug;39(3):384-9. doi: 10.3758/bf03193007. PMID 17958149
- [Background] Masyn KE. Discrete-Time Survival Factor Mixture Analysis for Low-Frequency Recurrent Event Histories. Res Hum Dev. 2009;6(2-3):165-194. doi: 10.1080/15427600902911270. PMID 24489519
- [Background] McCabe K, Yeh M. Parent-child interaction therapy for Mexican Americans: a randomized clinical trial. J Clin Child Adolesc Psychol. 2009 Sep;38(5):753-9. doi: 10.1080/15374410903103544. PMID 20183659
- [Background] McCanne TR, Hagstrom AH. Physiological hyperreactivity to stressors in physical child abusers and individuals at risk for being physically abusive. Aggression and Violent Behavior 1: 345-358, 1996.
- [Background] McDermott JM, Westerlund A, Zeanah CH, Nelson CA, Fox NA. Early adversity and neural correlates of executive function: implications for academic adjustment. Dev Cogn Neurosci. 2012 Feb 15;2 Suppl 1(Suppl 1):S59-66. doi: 10.1016/j.dcn.2011.09.008. Epub 2011 Oct 19. PMID 22682911
- [Background] Milner JS. The Child Abuse Potential Inventory MANUAL (2nd ed.). DeKalb, IL: Psytec, Inc., 1986.
- [Background] Milner JS. Assessing physical child abuse risk: The Child Abuse Potential Inventory. Clinical Psychology Review, 14, 547-583, 1994.
- [Background] Minuchin S. Families and family therapy. Oxford, England: Harvard University Press, 1974.
- [Background] Moadab I, Gilbert T, Dishion TJ, Tucker DM. Frontolimbic activity in a frustrating task: covariation between patterns of coping and individual differences in externalizing and internalizing symptoms. Dev Psychopathol. 2010 May;22(2):391-404. doi: 10.1017/S0954579410000131. PMID 20423549
- [Background] Moffitt T. The neuropsychology of conduct disorder. Development and Psychopathology 5: 135-151, 1993.
- [Background] Morgan-Lopez AA, MacKinnon DP. Demonstration and evaluation of a method for assessing mediated moderation. Behav Res Methods. 2006 Feb;38(1):77-87. doi: 10.3758/bf03192752. PMID 16817516
- [Background] Muller D, Judd CM, Yzerbyt VY. When moderation is mediated and mediation is moderated. J Pers Soc Psychol. 2005 Dec;89(6):852-63. doi: 10.1037/0022-3514.89.6.852. PMID 16393020
- [Background] Muthén BO, Curran PJ. General longitudinal modeling of individual differences in experimental designs: A latent variable framework for analysis and power estimation. Psychological Methods 2: 371-402, 1997.
- [Background] Muthén LK, Muthén BO. How to use a Monte Carlo study to decide on sample size and determine power. Structural Equation Modeling 9(4): 599-620, 2002.
- [Background] Muthén LK, Muthén BO. MPlus User's Guide (7th ed.). Los Angeles, CA: StatModel, 2012.
- [Background] National Scientific Council on the Developing Child. Excessive stress disrupts the architecture of the developing brain: Working Paper #3. Psychology & Health, 19, 237-246, 2005.
- [Background] Pandey AK, Kamarajan C, Tang Y, Chorlian DB, Roopesh BN, Manz N, Stimus A, Rangaswamy M, Porjesz B. Neurocognitive deficits in male alcoholics: an ERP/sLORETA analysis of the N2 component in an equal probability Go/NoGo task. Biol Psychol. 2012 Jan;89(1):170-82. doi: 10.1016/j.biopsycho.2011.10.009. Epub 2011 Oct 21. PMID 22024409
- [Background] Pine DS, Mogg K, Bradley BP, Montgomery L, Monk CS, McClure E, Guyer AE, Ernst M, Charney DS, Kaufman J. Attention bias to threat in maltreated children: implications for vulnerability to stress-related psychopathology. Am J Psychiatry. 2005 Feb;162(2):291-6. doi: 10.1176/appi.ajp.162.2.291. PMID 15677593
- [Background] Pine DS, Wasserman GA, Miller L, Coplan JD, Bagiella E, Kovelenku P, Myers MM, Sloan RP. Heart period variability and psychopathology in urban boys at risk for delinquency. Psychophysiology. 1998 Sep;35(5):521-9. doi: 10.1017/s0048577298970846. PMID 9715096
- [Background] Pollak SD. Mechanisms Linking Early Experience and the Emergence of Emotions: Illustrations From the Study of Maltreated Children. Curr Dir Psychol Sci. 2008 Dec;17(6):370-375. doi: 10.1111/j.1467-8721.2008.00608.x. PMID 21701602
- [Background] Pollak SD, Cicchetti D, Klorman R, Brumaghim JT. Cognitive Brain Event-Related Potentials and Emotion Processing in Maltreated Children. Child Dev. 1997 Oct;68(5):773-787. doi: 10.1111/j.1467-8624.1997.tb01961.x. PMID 29106724
- [Background] Pollak SD, Vardi S, Putzer Bechner AM, Curtin JJ. Physically abused children's regulation of attention in response to hostility. Child Dev. 2005 Sep-Oct;76(5):968-77. doi: 10.1111/j.1467-8624.2005.00890.x. PMID 16149995
- [Background] Ponitz CC, McClelland MM, Matthews JS, Morrison FJ. A structured observation of behavioral self-regulation and its contribution to kindergarten outcomes. Dev Psychol. 2009 May;45(3):605-19. doi: 10.1037/a0015365. PMID 19413419
- [Background] Porges SW. Orienting in a defensive world: mammalian modifications of our evolutionary heritage. A Polyvagal Theory. Psychophysiology. 1995 Jul;32(4):301-18. doi: 10.1111/j.1469-8986.1995.tb01213.x. PMID 7652107
- [Background] Porges SW. The polyvagal theory: phylogenetic substrates of a social nervous system. Int J Psychophysiol. 2001 Oct;42(2):123-46. doi: 10.1016/s0167-8760(01)00162-3. PMID 11587772
- [Background] Posne MI, Rothbart MK. Developing mechanisms of self-regulation. Dev Psychopathol. 2000 Summer;12(3):427-41. doi: 10.1017/s0954579400003096. PMID 11014746
- [Background] Preacher KJ, Hayes AF. Asymptotic and resampling strategies for assessing and comparing indirect effects in multiple mediator models. Behav Res Methods. 2008 Aug;40(3):879-91. doi: 10.3758/brm.40.3.879. PMID 18697684
- [Background] Pu J, Schmeichel BJ, Demaree HA. Cardiac vagal control predicts spontaneous regulation of negative emotional expression and subsequent cognitive performance. Biological Psychology 84: 531-540, 2010.
- [Background] Racer KH, Dishion TJ. Disordered Attention: Implications for Understanding and Treating Internalizing and Externalizing Disorders in Childhood. Cogn Behav Pract. 2012 Feb;19(1):31-40. doi: 10.1016/j.cbpra.2010.06.005. PMID 23365493
- [Background] Racer KH, Gilbert TT, Luu P, Felver-Gant J, Abdullaev Y, Dishion TJ. Attention network performance and psychopathic symptoms in early adolescence: an ERP study. J Abnorm Child Psychol. 2011 Oct;39(7):1001-12. doi: 10.1007/s10802-011-9522-6. PMID 21607659
- [Background] Repetti RL, Taylor SE, Seeman TE. Risky families: family social environments and the mental and physical health of offspring. Psychol Bull. 2002 Mar;128(2):330-66. PMID 11931522
- [Background] Reynolds CR, Kamphaus RW. Behavior assessment system for children (2nd ed.). Circle Pines, MN: American Guidance Service, 2004.
- [Background] Robins LN, Helzer JE, Croughan J, Ratcliff KS. National Institute of Mental Health Diagnostic Interview Schedule. Its history, characteristics, and validity. Arch Gen Psychiatry. 1981 Apr;38(4):381-9. doi: 10.1001/archpsyc.1981.01780290015001. PMID 6260053
- [Background] Rogosch FA, Cicchetti D, Aber JL. The role of child maltreatment in early deviations in cognitive and affective processing abilities and later peer relationship problems. Development and Psychopathology 7: 591-609, 1995.
- [Background] Roth RM, Isquith PK, Gioia GA. BRIEF-A: Behavior Rating Inventory of Executive Function-Adult Version. Lutz, FL: Psychological Assessment Resources, 2005.
- [Background] Rothbart MK, Ahadi SA, Evans DE. Temperament and personality: origins and outcomes. J Pers Soc Psychol. 2000 Jan;78(1):122-35. doi: 10.1037//0022-3514.78.1.122. PMID 10653510
- [Background] Sameroff AJ, Lewis M, Miller SM. Handbook of developmental psychopathology (2nd ed.). New York, NY: Kluwer Academic/Plenum Press, 2000.
- [Background] Sarason IG, Johnson JH, Siegel JM. Assessing the impact of life changes: development of the Life Experiences Survey. J Consult Clin Psychol. 1978 Oct;46(5):932-46. doi: 10.1037//0022-006x.46.5.932. No abstract available. PMID 701572
- [Background] Scaramella LV, Neppl TK, Ontai LL, Conger RD. Consequences of socioeconomic disadvantage across three generations: parenting behavior and child externalizing problems. J Fam Psychol. 2008 Oct;22(5):725-33. doi: 10.1037/a0013190. PMID 18855508
- [Background] Schafer JL, Graham JW. Missing data: our view of the state of the art. Psychol Methods. 2002 Jun;7(2):147-77. PMID 12090408
- [Background] Shackman JE, Shackman AJ, Pollak SD. Physical abuse amplifies attention to threat and increases anxiety in children. Emotion. 2007 Nov;7(4):838-52. doi: 10.1037/1528-3542.7.4.838. PMID 18039053
- [Background] Shonkoff JP, Fisher PA. Rethinking evidence-based practice and two-generation programs to create the future of early childhood policy. Dev Psychopathol. 2013 Nov;25(4 Pt 2):1635-53. doi: 10.1017/S0954579413000813. PMID 24342860
- [Background] Shonkoff JP, Garner AS; Committee on Psychosocial Aspects of Child and Family Health; Committee on Early Childhood, Adoption, and Dependent Care; Section on Developmental and Behavioral Pediatrics. The lifelong effects of early childhood adversity and toxic stress. Pediatrics. 2012 Jan;129(1):e232-46. doi: 10.1542/peds.2011-2663. Epub 2011 Dec 26. PMID 22201156
- [Background] Sinharay S, Stern HS, Russell D. The use of multiple imputation for the analysis of missing data. Psychol Methods. 2001 Dec;6(4):317-29. PMID 11778675
- [Background] Skowron EA. Parent differentiation of self and child competence in low-income, urban families. Journal of Counseling Psychology 52: 337-342, 2005.
- [Background] Skowron EA, Reinemann DHS. Psychological interventions for child maltreatment: A metaanalysis. Psychotherapy: Theory, Research, Practice, and Training 42: 52-71, 2005.
- [Background] Skowron EA, Cipriano-Essel E, Benjamin LS, Pincus AL, Van Ryzin MJ. Cardiac Vagal Tone and Quality of Parenting Show Concurrent and Time-Ordered Associations That Diverge in Abusive, Neglectful, and Non-Maltreating Mothers. Couple Family Psychol. 2013 Jun 1;2(2):95-115. doi: 10.1037/cfp0000005. PMID 24729945
- [Background] Skowron EA, Cipriano-Essel E, Gatzke-Kopp LM, Teti DM, Ammerman RT. Early adversity, RSA, and inhibitory control: evidence of children's neurobiological sensitivity to social context. Dev Psychobiol. 2014 Jul;56(5):964-78. doi: 10.1002/dev.21175. Epub 2013 Oct 19. PMID 24142832
- [Background] Skowron EA, Khurana A, Gatzke-Kopp L. (under review). Latent classes of dyadic rupture-repair processes predict children's RSA and inhibitory control.
- [Background] Skowron EA, Loken E, Gatzke-Kopp LM, Cipriano-Essel EA, Woehrle PL, Van Epps JJ, Gowda A, Ammerman RT. Mapping cardiac physiology and parenting processes in maltreating mother-child dyads. J Fam Psychol. 2011 Oct;25(5):663-74. doi: 10.1037/a0024528. PMID 21842991
- [Background] Smith TW, Cribbet MR, Nealey-Moore JB, Uchino BN, Williams PG, Mackenzie J, Thayer JF. Matters of the variable heart: respiratory sinus arrhythmia response to marital interaction and associations with marital quality. J Pers Soc Psychol. 2011 Jan;100(1):103-19. doi: 10.1037/a0021136. PMID 20954783
- [Background] Spanier GB. Measuring dyadic adjustment: New scales for assessing the quality of marriage and similar dyads. Journal of Marriage and the Family 47: 15-28, 1976.
- [Background] Straus MA, Hamby SL, Boney-McCoy S, Sugarman DB. The revised Conflict Tactics Scales (CTS2): Development and preliminary psychometric data. Journal of Family Issues 17: 283-316, 1996.
- [Background] Stroop JR. Studies of interference in serial verbal reactions. Journal of Experimental Psychology 18: 643-662, 1935.
- [Background] Suchman NE, Pajulo M, Mayes LC. (Eds.). Parenting and substance abuse: Developmental approaches to intervention. New York, NY: Oxford University Press, 2013.
- [Background] Tang YY, Ma Y, Wang J, Fan Y, Feng S, Lu Q, Yu Q, Sui D, Rothbart MK, Fan M, Posner MI. Short-term meditation training improves attention and self-regulation. Proc Natl Acad Sci U S A. 2007 Oct 23;104(43):17152-6. doi: 10.1073/pnas.0707678104. Epub 2007 Oct 11. PMID 17940025
- [Background] Tarullo AR, Gunnar MR. Child maltreatment and the developing HPA axis. Horm Behav. 2006 Nov;50(4):632-9. doi: 10.1016/j.yhbeh.2006.06.010. Epub 2006 Jul 28. PMID 16876168
- [Background] Thayer JF, Lane RD. A model of neurovisceral integration in emotion regulation and dysregulation. J Affect Disord. 2000 Dec;61(3):201-16. doi: 10.1016/s0165-0327(00)00338-4. PMID 11163422
- [Background] Trickett PK. Maladaptive development of school-aged, physically abused children: Relationships with the child-rearing context. Journal of Family Psychology 7: 134-147, 1993.
- [Background] Trocmé N. Development and preliminary evaluation of the Ontario Child Neglect Index. Child Maltreatment 1: 145-155, 1996.
- [Background] U.S. Department of Health and Human Services, Administration for Children and Families, Administration on Children, Youth and Families, Children's Bureau. Child Maltreatment 2011, 2012.
- [Background] Urquiza AJ, McNeil CB. Parent-Child Interaction Therapy: An intensive dyadic intervention for physically abusive families. Child Maltreatment 1: 134-144, 1996.
- [Background] van Noordt SJ, Segalowitz SJ. Performance monitoring and the medial prefrontal cortex: a review of individual differences and context effects as a window on self-regulation. Front Hum Neurosci. 2012 Jul 11;6:197. doi: 10.3389/fnhum.2012.00197. eCollection 2012. PMID 22798949
- [Background] Vanderwert RE, Marshall PJ, Nelson CA 3rd, Zeanah CH, Fox NA. Timing of intervention affects brain electrical activity in children exposed to severe psychosocial neglect. PLoS One. 2010 Jul 1;5(7):e11415. doi: 10.1371/journal.pone.0011415. PMID 20617175
- [Background] Walker S, O'Connor DB, Schaefer A. Brain potentials to emotional pictures are modulated by alexithymia during emotion regulation. Cogn Affect Behav Neurosci. 2011 Dec;11(4):463-75. doi: 10.3758/s13415-011-0042-1. PMID 21614450
- [Background] West RL, Hastings EC. Self-regulation and recall: growth curve modeling of intervention outcomes for older adults. Psychol Aging. 2011 Dec;26(4):803-12. doi: 10.1037/a0023784. Epub 2011 May 23. PMID 21604891
- [Background] Wilson SR, Rack JJ, Shi X, Norris AM. Comparing physically abusive, neglectful, and non-maltreating parents during interactions with their children: a meta-analysis of observational studies. Child Abuse Negl. 2008 Sep;32(9):897-911. doi: 10.1016/j.chiabu.2008.01.003. Epub 2008 Oct 23. PMID 18950859
- [Background] Woltering S, Granic I, Lamm C, Lewis MD. Neural changes associated with treatment outcome in children with externalizing problems. Biol Psychiatry. 2011 Nov 1;70(9):873-9. doi: 10.1016/j.biopsych.2011.05.029. Epub 2011 Jul 8. PMID 21741030
- [Background] Yu F, Yuan J, Luo YJ. Auditory-induced emotion modulates processes of response inhibition: an event-related potential study. Neuroreport. 2009 Jan 7;20(1):25-30. doi: 10.1097/WNR.0b013e32831ac9b1. PMID 18978645
- [Background] Zhou Q, Chen SH, Main A. Commonalities and differences in the research on children's effortful control and executive function: A call for an integrated model of self-regulation. Child Development Perspectives 6: 112-121, 2012.
- [Derived] Skowron EA, Nekkanti AK, Skoranski AM, Scholtes CM, Lyons ER, Mills KL, Bard D, Rock A, Berkman E, Bard E, Funderburk BW. Randomized trial of parent-child interaction therapy improves child-welfare parents' behavior, self-regulation, and self-perceptions. J Consult Clin Psychol. 2024 Feb;92(2):75-92. doi: 10.1037/ccp0000859. Epub 2023 Dec 7. PMID 38059943
- [Derived] Nekkanti AK, Jeffries R, Scholtes CM, Shimomaeda L, DeBow K, Norman Wells J, Lyons ER, Giuliano RJ, Gutierrez FJ, Woodlee KX, Funderburk BW, Skowron EA. Study Protocol: The Coaching Alternative Parenting Strategies (CAPS) Study of Parent-Child Interaction Therapy in Child Welfare Families. Front Psychiatry. 2020 Sep 2;11:839. doi: 10.3389/fpsyt.2020.00839. eCollection 2020. PMID 33101068

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Number Started represents the number of parent participants and the number of child participants. There were 204 parent participants and 204 child participants enrolled for a total of 408 participants (in 204 parent-child dyads).
Groups:
- Services As Usual (SAU): Participants receive all the usual services provided by DHS- Children's Services.
- Parent Child Interaction Therapy (PCIT): Participants receive Parent Child Interaction Therapy (PCIT). PCIT is designed to improve child functioning by interrupting patterns of harsh, coercive interaction and enhancing parents' warm, positive parenting, autonomy support, and competent child management skills.
  Parent Child Interaction Therapy: PCIT is a 16-20 session live-coaching parenting intervention. PCIT for Child Welfare families is delivered in two sequential treatment phases following a motivational enhancement training: Phase 1, Child-Directed Interaction (CDI) to enhance positive parenting and interrupt harsh aversive parenting, and Phase 2, Parent-Directed Interaction (PDI) to coach effective parent commands and a consistent time-out protocol when child disobeys.
Period: Overall Study
Arm/Group | Services As Usual (SAU) | Parent Child Interaction Therapy (PCIT)
Started | 168 ((84 parents and 84 children)) | 240 ((120 parents and 120 children))
Completed | 133 ((68 parents and 65 children)) | 193 ((100 parents and 93 children))
Not Completed | 35 | 47
Not completed — COVID-19 shutdown of lab | 4 | 6
Not completed — Lost to Follow-up | 31 | 41

BASELINE CHARACTERISTICS:
Population: Note the sample is comprised of N = 204 parent and child dyads or 408 total individuals. There are 84 parent-child dyads (168 total individuals) in the services-as-usual condition and 120 parent-child dyads (240 total individuals) in the PCIT intervention condition.
Groups:
- Parent Child Interaction Therapy (PCIT): Participants randomized to receive Parent Child Interaction Therapy (PCIT). PCIT is designed to improve child functioning by interrupting patterns of harsh, coercive interaction and enhancing parents' warm, positive parenting, autonomy support, and competent child management skills.
  Parent Child Interaction Therapy: PCIT is a 16-20 session live-coaching parenting intervention. PCIT for Child Welfare families is delivered in two sequential treatment phases following a motivational enhancement training: Phase 1, Child-Directed Interaction (CDI) to enhance positive parenting and interrupt harsh aversive parenting, and Phase 2, Parent-Directed Interaction (PDI) to coach effective parent commands and a consistent time-out protocol when child disobeys.
- Total: Total of all reporting groups
Arm/Group | Services As Usual (SAU) | Parent Child Interaction Therapy (PCIT) | Total
Number analyzed (Participants) | 168 | 240 | 408
Age, Continuous [Mean (Standard Deviation); unit: years] — This is PARENT age in years Population: Only the 204 parents' age data were included in this analysis.
  years
    number analyzed (Participants) | 84 | 120 | 204
    (all) | 32.12 (5.82) | 32.41 (6.70) | 32.29 (6.34)
Sex: Female, Male [Count of Participants; unit: Participants] — Parent Sex: Female, Male Population: Only PARENT sex is included in this analysis.
  Participants
    number analyzed (Participants) | 84 | 120 | 204
    Female | 73 | 107 | 180
    Male | 11 | 13 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: PARENT and CHILD data are reported in separate sections below.
  Participants
    PARENT participants: number analyzed (Participants) | 84 | 120 | 204
    PARENT participants: European American/White | 62 | 82 | 144
    PARENT participants: Multiracial/Multiethnic | 15 | 27 | 42
    PARENT participants: Hispanic American/Latinx | 2 | 3 | 5
    PARENT participants: African American/Black | 2 | 2 | 4
    PARENT participants: Asian/Pacific Islander | 0 | 3 | 3
    PARENT participants: Native American/Alaskan Aleutian | 2 | 1 | 3
    PARENT participants: Not reported | 1 | 2 | 3
    CHILD participants: number analyzed (Participants) | 84 | 120 | 204
    CHILD participants: European American/White | 49 | 68 | 117
    CHILD participants: Multiracial/Multiethnic | 27 | 46 | 73
    CHILD participants: Hispanic American/Latinx | 3 | 3 | 6
    CHILD participants: African American/Black | 2 | 1 | 3
    CHILD participants: Asian/Pacific Islander | 0 | 0 | 0
    CHILD participants: Native American/Alaskan Aleutian | 1 | 1 | 2
    CHILD participants: Not reported | 2 | 1 | 3
Participating child age (years) [Mean (Standard Deviation); unit: years] — Population: Only the CHILD participants' ages were included in this analysis.
  years
    number analyzed (Participants) | 84 | 120 | 204
    (all) | 4.8 (1.4) | 4.7 (1.4) | 4.8 (1.4)
Participating child sex [Count of Participants; unit: Participants] — Population: Only CHILD sex is included in this analysis.
  Participants
    number analyzed (Participants) | 84 | 120 | 204
    Male children | 50 | 62 | 112
    Female children | 34 | 58 | 92
Parent education [Count of Participants; unit: Participants] — Population: Only PARENT education levels are included in this analysis.
  Participants
    number analyzed (Participants) | 84 | 120 | 204
    Less than high school education | 14 | 20 | 34
    High school education | 43 | 58 | 101
    Post-high school education | 27 | 42 | 69
Marital status [Count of Participants; unit: Participants] — Population: Only PARENT marital status is included here.
  Participants
    number analyzed (Participants) | 84 | 120 | 204
    Single | 64 | 74 | 138
    Married or living together | 20 | 46 | 66

OUTCOME MEASURES:

1. Primary Outcome: DPICS-IV Observed Parenting Skills (During Child-Led Play)
Description: Dyadic Parent-Child Interaction Coding System (DPICS) coded positive "PRIDE" parenting skills and negative "Don't skills" parenting behaviors during the DPICS Child-Led Play task. Scores reflect behavioral counts during the 5-minute task, with higher scores reflecting more behaviors. Higher positive parenting scores reflect better outcomes, whereas higher negative parenting scores reflect worse outcomes.
Time Frame: Pre- and Post-intervention (8 months)
Population: These participating child welfare-involved families were block-randomized to condition by child sex and age, with allocation ratio of PCIT to control group conditions at 1.5:1 to ensure that a sufficient number of families accessed the intervention.
Measure: Mean (Standard Deviation); unit: number of behaviors
Groups:
- Parent Child Interaction Therapy (PCIT): All participants randomized to PCIT condition.
  Participants receive Parent Child Interaction Therapy (PCIT). PCIT is designed to improve child functioning by interrupting patterns of harsh, coercive interaction and enhancing parents' warm, positive parenting, autonomy support, and competent child management skills.
  Parent Child Interaction Therapy: PCIT is a 16-20 session live-coaching parenting intervention. PCIT for Child Welfare families is delivered in two sequential treatment phases following a motivational enhancement training: Phase 1, Child-Directed Interaction (CDI) to enhance positive parenting and interrupt harsh aversive parenting, and Phase 2, Parent-Directed Interaction (PDI) to coach effective parent commands and a consistent time-out protocol when child disobeys.
- Parent Child Interaction Therapy (PCIT) (Engagers Only): All participants randomized to PCIT condition who engaged in 1+ sessions.
  Participants receive Parent Child Interaction Therapy (PCIT). PCIT is designed to improve child functioning by interrupting patterns of harsh, coercive interaction and enhancing parents' warm, positive parenting, autonomy support, and competent child management skills.
  Parent Child Interaction Therapy: PCIT is a 16-20 session live-coaching parenting intervention. PCIT for Child Welfare families is delivered in two sequential treatment phases following a motivational enhancement training: Phase 1, Child-Directed Interaction (CDI) to enhance positive parenting and interrupt harsh aversive parenting, and Phase 2, Parent-Directed Interaction (PDI) to coach effective parent commands and a consistent time-out protocol when child disobeys.
Arm/Group | Services As Usual (SAU) | Parent Child Interaction Therapy (PCIT) | Parent Child Interaction Therapy (PCIT) (Engagers Only)
Number analyzed (Participants) | 84 | 120 | 79
number of behaviors
  Positive Parenting "PRIDE" skills (pre-treatment) | 2.32 (2.32) | 2.63 (2.92) | 2.86 (3.10)
  Positive Parenting "PRIDE" skills (post-treatment) | 2.11 (2.20) | 8.01 (9.61) | 10.19 (10.47)
  Negative Parenting "Don't" skills (pre-treatment) | 23.62 (11.66) | 23.61 (11.78) | 24.16 (11.92)
  Negative Parenting "Don't" skills (post-treatment) | 21.80 (11.31) | 14.82 (9.99) | 13.30 (9.42)

2. Primary Outcome: DPICS-IV Observational Coding During Clean Up Situation Task
Description: DPICS-Coded Positive "PRIDE" Parenting skills, Effective Parent Commands, and Child Compliance behaviors during the DPICS Clean Up Situation task. Positive parenting scores reflect the percentage of total coded behaviors during the task that are positive "PRIDE" skills. Effective (direct) parent commands reflect the percentage of all commands that were direct, compliable commands. Child compliance scores reflected the percentage of effective, direct commands that child complied with in the immediately following behavioral turn. High scores on all three scales reflect better outcomes.
Time Frame: Pre- and Post-intervention (8 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of all parenting behaviors
Arm/Group | Services As Usual (SAU) | Parent Child Interaction Therapy (PCIT) | Parent Child Interaction Therapy (PCIT) (Engagers Only)
Number analyzed (Participants) | 84 | 120 | 79
percentage of all parenting behaviors
  Effective commands (pre-treatment) | 0.56 (0.26) | 0.54 (0.25) | 0.53 (0.24)
  Effective commands (post-treatment) | 0.63 (0.27) | 0.60 (0.29) | 0.59 (0.29)
  Child compliance with parent commands (pre-treatment) | 0.69 (0.28) | 0.73 (0.28) | 0.71 (0.31)
  Child compliance with parent commands (post-treatment) | 0.78 (0.22) | 0.76 (0.29) | 0.75 (0.31)
  Positive Parenting "PRIDE" skills (pre-treatment) | 0.65 (0.27) | 0.62 (0.29) | 0.63 (0.28)
  Positive Parenting "PRIDE" skills (post-treatment) | 0.69 (0.28) | 0.70 (0.31) | 0.71 (0.31)

3. Primary Outcome: Stop Signal Task: Increased Parent Inhibitory Control
Description: The Stop Signal Response Time (SSRT) was used to assess the efficiency of parent inhibitory control process or time in milliseconds needed to engage an inhibitory response. Lower SSRT scores reflect faster reaction times and better inhibitory control.
Time Frame: pre- and post-intervention (8 months)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Services As Usual (SAU) | Parent Child Interaction Therapy (PCIT) | Parent Child Interaction Therapy (PCIT) (Engagers Only)
Number analyzed (Participants) | 84 | 120 | 79
milliseconds
  Stop signal response time (SSRT) (pre-treatment) | 252.84 (68.07) | 248.25 (54.40) | 251.44 (58.18)
  Stop signal response time (SSRT) (post-treatment) | 255.16 (57.94) | 237.45 (47.89) | 236.28 (45.33)

4. Secondary Outcome: Reduced Child Maltreatment (CM) Recidivism
Description: Fewer new episodes of CM per Maltreatment Classification Coding of Child Welfare case records
Time Frame: up to 1 year posttreatment
Population: These data are not available from DHS child welfare on the study participants and thus not available to our study team to report here. We have been told that this is due to the fact that the DHS agency internal record-keeping systems do not have data on the study families.
Groups:
- Parent Child Interaction Therapy (PCIT): Participants receive Parent Child Interaction Therapy (PCIT). PCIT is designed to improve child functioning by interrupting patterns of harsh, coercive interaction and enhancing parents' warm, positive parenting, autonomy support, and competent child management skills.
  .
  Parent Child Interaction Therapy: PCIT is a 16-20 session live-coaching parenting intervention. PCIT for Child Welfare families is delivered in two sequential treatment phases following a motivational enhancement training: Phase 1, Child-Directed Interaction (CDI) to enhance positive parenting and interrupt harsh aversive parenting, and Phase 2, Parent-Directed Interaction (PDI) to coach effective parent commands and a consistent time-out protocol when child disobeys.
Arm/Group | Services As Usual (SAU) | Parent Child Interaction Therapy (PCIT)
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: BRIEF-A: Emotional Control Scale (Increased Parent Emotion Regulation)
Description: Parents self-report on the BRIEF- A Emotional Control problem scale, with lower scores reflecting fewer emotion control problems (i.e., better emotion regulation). Standardized T-scores (M=50, SD = 10) are obtained.
Time Frame: pre- and post-intervention (8 months)
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Services As Usual (SAU) | Parent Child Interaction Therapy (PCIT) | Parent Child Interaction Therapy (PCIT) (Engagers Only)
Number analyzed (Participants) | 84 | 120 | 79
T-scores
  Emotional Control problems (pre-treatment) | 52.57 (9.18) | 53.95 (10.87) | 55.06 (11.38)
  Emotional Control problems (post-treatment) | 54.95 (11.21) | 52.72 (11.03) | 53.33 (10.97)

6. Other Pre Specified Outcome: BRIEF (Behavioral Rating Inventory of Executive Function) Children's Outcomes
Description: Children's BRIEF scores per parent-report on Inhibit, Shift, and Emotional Control problems scales, with lower scores reflecting fewer regulatory problems. Standardized T-scores (M=50, SD = 10) are obtained.
Time Frame: pre- and post-intervention
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Services As Usual (SAU) | Parent Child Interaction Therapy (PCIT) | Parent Child Interaction Therapy (PCIT) (Engagers Only)
Number analyzed (Participants) | 84 | 120 | 79
T-scores
  Inhibition problems (pre-treatment) | 59.11 (12.00) | 58.36 (12.34) | 59.84 (11.76)
  Inhibition problems (post-treatment) | 60.12 (11.72) | 57.98 (10.88) | 58.55 (10.92)
  Shift problems (pretreatment) | 54.86 (13.08) | 57.10 (11.55) | 58.63 (11.07)
  Shift problems (posttreatment) | 55.46 (12.95) | 55.27 (10.89) | 55.90 (10.94)
  Emotional control problems (pretreatment) | 54.30 (12.58) | 54.79 (11.76) | 56.09 (12.07)
  Emotional control problems (posttreatment) | 54.42 (10.30) | 52.87 (11.14) | 53.03 (11.49)

7. Other Pre Specified Outcome: Parent Physiological Regulation
Description: physiological regulation (Respiratory Sinus Arrhythmia or RSA scores, are a peripheral physiological marker of emotion regulation reflecting parents' parasympathetic nervous system linked cardiac activity. RSA scores were obtained from parents at rest and in response to emotionally salient interactions with their child. Higher RSA scores reflect greater parasympathetic cardiac regulation (better outcome).
Time Frame: pre- and post-intervention
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Services As Usual (SAU) | Parent Child Interaction Therapy (PCIT) | Parent Child Interaction Therapy (PCIT) (Engagers Only)
Number analyzed (Participants) | 84 | 120 | 79
ms^2
  Parent Resting RSA (at pretreatment) | 6.30 (1.38) | 5.97 (1.45) | 5.88 (1.53)
  Parent Resting RSA (at posttreatment) | 5.77 (1.59) | 5.57 (1.71) | 5.35 (1.71)
  Parent RSA during DPICS Child-Led Play Task (pretreatment) | 5.99 (1.38) | 5.76 (1.37) | 5.67 (1.44)
  Parent RSA during DPICS Child-Led Play Task (posttreatment) | 5.57 (1.48) | 5.58 (1.54) | 5.52 (1.57)
  Parent RSA during DPICS Clean Up Task (pretreatment) | 6.05 (1.22) | 5.79 (1.29) | 5.71 (1.32)
  Parent RSA during DPICS Clean Up Task (posttreatment) | 5.81 (1.44) | 5.51 (1.39) | 5.41 (1.43)
  Parent RSA during Social Engagement task (pretreatment) | 6.51 (1.24) | 6.19 (1.36) | 6.02 (1.43)
  Parent RSA during Social Engagement task (posttreatment) | 6.27 (1.48) | 5.98 (1.46) | 5.85 (1.47)

8. Other Pre Specified Outcome: Child Emotion Regulation
Description: Emotional go/no-go task performance: False alarms to anger. Higher scores reflect greater rate of false alarms to anger (worse outcome).
Time Frame: Post intervention (6 mo)
Measure: Mean (Standard Deviation); unit: percentage of responses
Arm/Group | Services As Usual (SAU) | Parent Child Interaction Therapy (PCIT) | Parent Child Interaction Therapy (PCIT) (Engagers Only)
Number analyzed (Participants) | 84 | 120 | 79
percentage of responses
  Child False Alarms to Anger (pretreatment) | 0.38 (0.27) | 0.40 (0.31) | 0.41 (0.31)
  Child False Alarms to Anger (posttreatment) | 0.38 (0.28) | 0.34 (0.24) | 0.35 (0.24)

9. Other Pre Specified Outcome: Child Physiological Regulation
Description: physiological regulation (Respiratory Sinus Arrhythmia or RSA scores, are a peripheral physiological marker of emotion regulation reflecting children's parasympathetic nervous system linked cardiac activity. RSA scores were obtained from children at rest and in response to emotionally salient interactions with their parent. Higher RSA scores reflect greater parasympathetic cardiac regulation (better outcome).
Time Frame: pre- and post-intervention (8 months)
Population: CHILD RSA data reported here
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Services As Usual (SAU) | Parent Child Interaction Therapy (PCIT) | Parent Child Interaction Therapy (PCIT) (Engagers Only)
Number analyzed (Participants) | 84 | 120 | 79
ms^2
  Child resting RSA (pretreatment) | 6.68 (1.20) | 6.41 (1.40) | 6.48 (1.34)
  Child resting RSA (postreatment) | 6.36 (1.33) | 6.47 (1.31) | 6.35 (1.25)
  Child RSA during child-led play task (pretreatment) | 5.40 (1.10) | 5.38 (1.10) | 5.42 (1.12)
  Child RSA during child-led play task (posttreatment) | 5.28 (1.04) | 5.33 (1.22) | 5.29 (1.18)
  Child RSA during clean-up task (pretreatment) | 4.95 (0.96) | 4.92 (1.05) | 4.98 (1.07)
  Child RSA during clean-up task (postreatment) | 4.73 (1.18) | 4.79 (1.22) | 4.67 (1.21)
  Child RSA during Social Engagement task with parent (pretreatment) | 6.10 (1.14) | 5.95 (1.23) | 5.98 (1.23)
  Child RSA during Social Engagement task with parent (postreatment) | 5.91 (1.11) | 6.05 (1.11) | 5.96 (1.09)

10. Other Pre Specified Outcome: Decreased Child Symptoms
Description: Trauma Symptom Checklist scores (TSCL-YC); T-scores are reported, in which 50 indicates the population mean with a standard deviation of 10; higher scores indicate greater trauma symptoms. Clinically significant elevations on the TSCL-YC are reflected by scores at or above T=70 cutoff
Time Frame: pre- and post-intervention (8 months)
Population: These are CHILD scores.
Measure: Mean (Standard Deviation); unit: t-scores
Arm/Group | Services As Usual (SAU) | Parent Child Interaction Therapy (PCIT) | Parent Child Interaction Therapy (PCIT) (Engagers Only)
Number analyzed (Participants) | 84 | 120 | 79
t-scores
  PTS-Arousal (pre-treatment) | 58.80 (13.74) | 59.70 (14.34) | 61.51 (14.72)
  PTS-Arousal (post-treatment) | 58.35 (14.17) | 57.05 (13.51) | 57.32 (13.83)
  PTS-Avoidance (pre-treatment) | 57.08 (15.33) | 59.04 (18.55) | 60.94 (19.05)
  PTS-Avoidance (post-treatment) | 56.96 (15.93) | 55.97 (16.63) | 57.84 (18.18)
  PTS-Intrusion (pre-treatment) | 57.47 (14.62) | 58.98 (16.98) | 61.65 (17.52)
  PTS-Intrusion (post-treatment) | 53.95 (10.83) | 56.00 (14.12) | 57.81 (15.75)
  Anxiety (pre-treatment) | 55.33 (10.59) | 59.25 (14.50) | 60.96 (14.10)
  Anxiety (post-treatment) | 54.23 (9.55) | 57.92 (14.50) | 58.78 (14.53)

11. Other Pre Specified Outcome: Eyberg Child Behavior Inventory (ECBI) Child Behavior Problem Scores (Decreased Disruptive Behavior Problems)
Description: The ECBI is comprised of parent-reported intensity of problem child behaviors (ECBI-Intensity score) and number of problem child behaviors (EBCI-Problem score). Standardized T-scores (M=50, SD=10) are reported, with lower scores reflecting more successful outcome.
Time Frame: pre- and post-intervention (8 months)
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Services As Usual (SAU) | Parent Child Interaction Therapy (PCIT) | Parent Child Interaction Therapy (PCIT) (Engagers Only)
Number analyzed (Participants) | 84 | 120 | 79
T-scores
  ECBI-Intensity child behavior problems (pre-treatment) | 58.61 (10.79) | 56.33 (10.38) | 57.56 (10.65)
  ECBI-Intensity child behavior problems (post-treatment) | 57.01 (9.31) | 51.35 (9.85) | 50.39 (9.94)
  ECBI-Number child behavior problems (pre-treatment) | 58.64 (11.79) | 55.74 (11.08) | 57.00 (11.46)
  ECBI-Number child behavior problems (post-treatment) | 56.13 (10.95) | 50.43 (9.67) | 50.46 (9.93)

12. Other Pre Specified Outcome: BRIEF-A: Parent Self-ratings
Description: Parents self-report on the BRIEF- A with lower scores reflecting fewer regulatory control problems. Standardized T-scores (M=50, SD = 10) are obtained.
Time Frame: pre- and post-intervention (8 months)
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Services As Usual (SAU) | Parent Child Interaction Therapy (PCIT) | Parent Child Interaction Therapy (PCIT) (Engagers Only)
Number analyzed (Participants) | 84 | 120 | 79
T-scores
  Emotional control problems (pretreatment) | 52.57 (9.18) | 53.95 (10.87) | 55.06 (11.38)
  Emotional control problems (posttreatment) | 54.95 (11.21) | 52.72 (11.03) | 53.33 (10.97)
  Inhibition problems (pre-treatment) | 55.15 (10.27) | 55.92 (9.93) | 55.95 (9.87)
  Inhibition problems (post-treatment) | 55.32 (9.99) | 54.41 (9.81) | 54.33 (9.74)
  Initiate problems (pre) | 52.50 (10.87) | 54.33 (10.95) | 54.51 (10.63)
  Initiate problems (post) | 53.83 (12.46) | 52.18 (10.97) | 52.93 (10.85)
  Monitor problems (pretreatment) | 50.93 (10.10) | 52.48 (10.06) | 53.19 (10.57)
  Monitor problems (posttreatment) | 52.24 (11.27) | 51.35 (9.85) | 51.46 (9.53)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the time frame encompassing data collection, from participant study entry through study completion, an average of 8 months.
Description: Our definition of adverse event is consistent with clinicaltrials.gov, and is "an untoward or unfavorable medical occurrence in a study participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research." No adverse events occurred in this study.
Groups:
- Services As Usual (SAU) - Parents; Services As Usual (SAU) - Children: Participants receive all the usual services provided by DHS- Children's Services.
- Parent Child Interaction Therapy (PCIT) - Parents; Parent Child Interaction Therapy (PCIT) - Children: Participants randomized to receive Parent Child Interaction Therapy (PCIT). PCIT is designed to improve child functioning by interrupting patterns of harsh, coercive interaction and enhancing parents' warm, positive parenting, autonomy support, and competent child management skills.
  Parent Child Interaction Therapy: PCIT is a 16-20 session live-coaching parenting intervention. PCIT for Child Welfare families is delivered in two sequential treatment phases following a motivational enhancement training: Phase 1, Child-Directed Interaction (CDI) to enhance positive parenting and interrupt harsh aversive parenting, and Phase 2, Parent-Directed Interaction (PDI) to coach effective parent commands and a consistent time-out protocol when child disobeys.
- Parent-Child Interaction Therapy (PCIT) Engagers Only - Parents; Parent-Child Interaction Therapy (PCIT) Engagers Only - Children: All participants randomized to PCIT condition who engaged in 1+ sessions.
Arm/Group | Services As Usual (SAU) - Parents | Services As Usual (SAU) - Children | Parent Child Interaction Therapy (PCIT) - Parents | Parent Child Interaction Therapy (PCIT) - Children | Parent-Child Interaction Therapy (PCIT) Engagers Only - Parents | Parent-Child Interaction Therapy (PCIT) Engagers Only - Children
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/84 | 0/120 | 0/120 | 0/79 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/84 | 0/120 | 0/120 | 0/79 | 0/79
Other Adverse Events (participants affected / at risk) | 0/84 | 0/84 | 0/120 | 0/120 | 0/79 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT02684903/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT02684903/SAP_001.pdf